CLINICAL TRIAL: NCT03830775
Title: A Prospective Randomized Double Blinded Controlled Trial of Non-Operative Management of TFCC Injuries
Acronym: TFCC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn as researcher left
Sponsor: Edna Rath (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Edna Rath, Human Protection Director, William Beaumont Army Medical Center
Organization: William Beaumont Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: williamBAMC
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Wrist Injuries; PRP
Keywords: TFCC; PRP
MeSH Terms: conditions — Wrist Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental - PRP injection (Experimental): 2cc of PRP is injected into the ulnocarpal joint
  Interventions: Procedure: Platelet-rich plasma (PRP)
- control - Saline injection (Placebo Comparator): 2cc of 0.9% sterile saline is injected into the ulnocarpal joint
  Interventions: Procedure: Platelet-rich plasma (PRP)

INTERVENTIONS:
Procedure: Platelet-rich plasma (PRP) — PRP is obtained from obtaining an autologous blood sample, which is then condensed in a small commercial centrifuge to isolate a concentrated sample of platelets and growth factors. This sample contains high concentrations of Platelet-derived growth factors (PDGF), transforming growth factors β (TGFβ), insulin-like growth factor-1 (IGF1), and vascular endothelial growth factor-1 (VEGF) all of which aid in healing of soft tissues. (Padilla) The blood sample is autologous, the concentration is prepared in the clinic, and the complications of the injection are no greater than any other injection given in the clinic.
  All patients will have a blood sample prepared for PRP. The patient will then be blinded and half will randomly be assigned to PRP injection (2cc) and half will be randomly assigned to placebo (2cc of 0.9% sterile saline)

SUMMARY:
Platelet-rich Plasma (PRP) is formed when a patient's blood sample is concentrated by a commercially available centrifuge. The sample then contains a high concentration of growth factors and has been used for numerous indications in a number of joints. This process has not yet been proven for non-operative management of the Triangular FibroCartilage Complex (TFCC), which is a very commonly injured soft tissue structure in the wrist. This study seeks to determine the efficacy of PRP for TFCC injuries.

DETAILED DESCRIPTION:
Platelet-rich Plasma (PRP) therapy has recently been indicated in the treatment of joint pain, arthritis, tendonitis, and to augment surgical treatment has become increasingly common (Hsu) PRP is obtained from obtaining an autologous blood sample, which is then condensed in a small commercial centrifuge to isolate a concentrated sample of platelets and growth factors. This sample contains high concentrations of Platelet-derived growth factors (PDGF), transforming growth factors β (TGFβ), insulin-like growth factor-1 (IGF1), and vascular endothelial growth factor-1 (VEGF) all of which aid in healing of soft tissues. (Padilla) The blood sample is autologous, the concentration is prepared in the clinic, and the complications of the injection are no greater than any other injection given in the clinic. (Hsu) In addition to being safe, PRP is efficacious. PRP has been well-studied including 10 prospective randomized controlled trials proving the effectiveness of PRP for knee osteoarthritis alone. (Dai) Strong evidence has also been reported in support of PRP use for bone healing (Bibbo, Tsai) tendinopathy (Mishra, Peerbooms) cartilage healing (Mei-Dan), and for augmentation of both ligament reconstruction (Fallouh) and repair (Mazzocca). Furthermore, the use of PRP has been shown to be a more cost effective treatment as compared to traditional methods in both chronic wound management and tendonitis (Gosens, Dougherty) PRP has not been studied in the wrist. Ulnar-sided wrist pain, most commonly involving the Triangular fibrocartilage complex (TFCC) is both difficult to diagnosis and treat,(Kleinmann, Fulcher, Graham) The TFCC is a meniscal homologue which acts to stabilize the wrist and to dissipate compressive forces. Tears within this soft tissue structure are painful and heal slowly. (Palmer, Palmer). Immobilization, steroid injections, or surgical treatment are the mainstays of treatment. However, PRP has not been studied as a treatment modality.

The purpose of this analysis is to study the efficacy of PRP injection in the treatment of a TFCC tear.

The null hypothesis is that there is no difference between injection into the wrist of PRP and saline (placebo).

The investigators hypothesize that PRP will reduce pain as compared to placebo.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients consenting for wrist injection, who additionally consent to participate in this study.
2. MRI which indicates a TFCC tear or Scapho-lunate ligament tear (SL)

Exclusion criteria:

1. Patients who do not choose to participate in the study or who do not wish to have an injection
2. Patients who want an injection - but do not want to be randomized.
3. Patients who do not complete one of the follow up documentations.
4. Patients who would like to know their injection (unblinded) may be informed but the investigators will still attempt to collect data as per protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Disability of the Army Shoulder Hand (DASH) | Pre-injection
  SCALE: 0-100 (0 being a good result and 100 being complete disability)
Disability of the Army Shoulder Hand (DASH) | 2 weeks post injection
  SCALE: 0-100 (0 being a good result and 100 being complete disability)
Disability of the Army Shoulder Hand (DASH) | 3 months post injection
  SCALE: 0-100 (0 being a good result and 100 being complete disability)
Disability of the Army Shoulder Hand (DASH) | 6 months post injection
  SCALE: 0-100 (0 being a good result and 100 being complete disability)
Disability of the Army Shoulder Hand (DASH) | 12 months post injection
  SCALE: 0-100 (0 being a good result and 100 being complete disability)

SECONDARY OUTCOMES:
Michigan Hand Outcome Questionnaire (MHOQ | Pre-injection, 2 weeks, 3 months
  SCALE: 0-100 (with 100 being a great result and 0 being considerable pain and dysfunction)
Mayo Wrist Score (Mayo) | Pre-injection, 2 weeks, 3 months, 6 months, 12 months
  SCALE: 0-100 (with 100 being a great result and 0 being considerable pain and dysfunction)
Pain Anxiety Symptom Scale (PASS) | Pre-injection, 2 weeks, 3 months
  SCALE: 0-100 (100 meaning a patient has a high level of anxiety, pain, apprehension; while a lower scale indicates a patient has no concerns or anxiety about pain. The average is about 38 and the standard deviation is 20)
Single Assessment Numerical Evaluation (SANE) | Pre-injection, 2 weeks, 3 months, 6 months, 12 months
  SCALE: 0-100 (with 100 being a great result and 0 being considerable pain and dysfunction)

CONTACTS AND LOCATIONS:
Overall Officials: John C Dunn, Principal Investigator — WBAMC Staff Hand Surgeon
Locations (1):
- Lola Norton, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padilla S, Orive G, Sanchez M, Anitua E, Hsu WK. Platelet-rich plasma in orthopaedic applications: evidence-based recommendations for treatment. J Am Acad Orthop Surg. 2014 Aug;22(8):469-70. doi: 10.5435/JAAOS-22-08-469. No abstract available. PMID 25063744
- [Background] Hsu WK, Mishra A, Rodeo SR, Fu F, Terry MA, Randelli P, Canale ST, Kelly FB. Platelet-rich plasma in orthopaedic applications: evidence-based recommendations for treatment. J Am Acad Orthop Surg. 2013 Dec;21(12):739-48. doi: 10.5435/JAAOS-21-12-739. PMID 24292930
- [Background] Dai WL, Zhou AG, Zhang H, Zhang J. Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2017 Mar;33(3):659-670.e1. doi: 10.1016/j.arthro.2016.09.024. Epub 2016 Dec 22. PMID 28012636
- [Background] Gosens T, Peerbooms JC, van Laar W, den Oudsten BL. Ongoing positive effect of platelet-rich plasma versus corticosteroid injection in lateral epicondylitis: a double-blind randomized controlled trial with 2-year follow-up. Am J Sports Med. 2011 Jun;39(6):1200-8. doi: 10.1177/0363546510397173. Epub 2011 Mar 21. PMID 21422467
- [Background] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Background] Palmer AK, Werner FW. The triangular fibrocartilage complex of the wrist--anatomy and function. J Hand Surg Am. 1981 Mar;6(2):153-62. doi: 10.1016/s0363-5023(81)80170-0. PMID 7229292
- [Background] Heyworth BE, Lee JH, Kim PD, Lipton CB, Strauch RJ, Rosenwasser MP. Hylan versus corticosteroid versus placebo for treatment of basal joint arthritis: a prospective, randomized, double-blinded clinical trial. J Hand Surg Am. 2008 Jan;33(1):40-8. doi: 10.1016/j.jhsa.2007.10.009. PMID 18261664